CLINICAL TRIAL: NCT03628209
Title: A Phase Ib/II Study to Evaluate the Safety, Feasibility and Efficacy of Nivolumab or Nivolumab in Combination With Azacitidine in Patients With Recurrent, Resectable Osteosarcoma
Brief Title: Nivolumab or Nivolumab and Azacitidine in Patients With Recurrent, Resectable Osteosarcoma
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-19487; CA209-9WW (Other: Bristol-Myers Squibb Protocol #)
Record Dates: First submitted 2018-08-08; First posted 2018-08-14 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Osteosarcoma; Osteosarcoma in Children; Osteosarcoma Recurrent; Sarcoma
Keywords: resectable osteosarcoma
MeSH Terms: conditions — Osteosarcoma; Sarcoma | interventions — Nivolumab; Azacitidine; Standard of Care

STUDY DESIGN:
Intervention Model Description: Phase Ib lead-in with extension to Phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation, Resection, Dose Expansion (Experimental): Participants will receive 1 cycle of neoadjuvant Nivolumab or Nivolumab + Azacitidine, followed by surgery to render them in surgical remission. Subsequently they will continue to receive Nivolumab or Nivolumab + Azacitidine for 12 additional cycles or until recurrence, whichever occurs first. Once the recommended Phase II dose (RP2D) is identified during Phase I, the Dose Expansion Phase II will be opened at this dose level. The Phase II portion of the study will consist of a maximum 33 evaluable patients (27-30 in addition to the 3-6 enrolled at RP2D on the Phase I portion).
  Interventions: Drug: Nivolumab; Drug: Azacitidine; Procedure: Post Treatment Surgery

INTERVENTIONS:
Drug: Nivolumab — Participants will be treated with Nivolumab intravenously (IV), 3 mg/kg on days 1 and 15 of each cycle.
  Other Names: Opdivo®
Drug: Azacitidine — Phase I Dose Escalation - Dose level 1: NA. Dose level 2: 60 mg/m^2. Dose level 3: 75 mg/m^2. Phase II Expansion - Treated at recommended Phase II dose (RP2D).
  Other Names: Vidaza®
Procedure: Post Treatment Surgery — Resection surgery at end of Cycle 1 treatment, day 28-35.
  Other Names: Standard of Care; Resection of disease

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of nivolumab, or nivolumab in combination with azacitidine in participants with recurrent, resectable osteosarcoma

DETAILED DESCRIPTION:
Treatment will be administered in 28 day cycles with the first cycle in the neoadjuvant setting. This will be followed by surgery to render the participant in surgical remission. Subsequently the participant will continue to receive treatment for up to 12 additional cycles or until recurrence, whichever occurs first. For participants with known bilateral lung recurrence, the nodule[s] in one lung should be resected, prior to the first cycle of chemotherapy. This trial was initially designed as a Phase 1/2 study; However, phase 2 will not proceed.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have had a histologic diagnosis of osteosarcoma at original diagnosis
* Disease Status: Patients with an isolated pulmonary recurrence of osteosarcoma can be enrolled on this study.

  * Any history of metastatic disease at a site other than lung would make the patient ineligible for this study.
  * The patient's treating team must consider the patient's disease to be resectable and the patient must be willing to undergo resection of all disease, including any lung lesion meeting criteria for likely metastatic disease, defined as: 3 or more lesions ≥ 3 mm in diameter OR a single lesion ≥ 5 mm.
  * Patients with bilateral disease are eligible provided their disease is considered resectable. Resectable pulmonary nodules are defined as nodules that can be removed without performing a pneumonectomy (e.g., nodules immediately adjacent to the main stem bronchus or main pulmonary vessels).
* Must have a performance status corresponding to Eastern Cooperative Oncology Group (ECOG) scores of 0, 1 or 2, using the Karnofsky scale for patients > 16 years of age and the Lansky scale for patients ≤ 16 years of age
* Prior Therapy: Participants must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to the start of protocol therapy.
* Participants must have normal organ and marrow function within 7 days of starting protocol therapy
* All participants and/or their parents or legal guardians must have the ability to understand and the willingness to sign a written informed consent/assent document
* Additional criteria may apply

Exclusion Criteria:

* Pregnancy or Breast Feeding
* Males and females of reproductive potential may not participate unless they have agreed to the use of, at minimum, two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective as outlined in study protocol documentation
* Concomitant Medications: Patients receiving the following are not eligible:

  * Corticosteroids or other immunosuppressive medications
* Patients who are currently receiving other investigational agents or other anti-cancer therapy
* Intercurrent Illnesses: Patients with uncontrolled intercurrent illness including, but not limited to:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness/social situations that would limit compliance with study requirements
* Autoimmune disorders: Patients with a history of any Grade autoimmune disorder are not eligible.
* Asymptomatic laboratory abnormalities (e.g., ANA, rheumatoid factor, altered thyroid function studies) will not render a patient ineligible in the absence of a diagnosis of an autoimmune disorder.
* Patients with ≥ Grade 2 hypothyroidism due to history of autoimmunity are not eligible. Note: Hypothyroidism due to previous irradiation or thyroidectomy will not impact eligibility
* Allergies: Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Nivolumab (e.g., another humanized antibody) or Azacitidine are not eligible
* Safety and Monitoring: Patients who are considered unable to comply with the safety monitoring requirements of the study are not eligible
* Patients with known HIV or hepatitis B or C are excluded
* Patients who have received prior solid organ transplantation are not eligible
* Patients who have received prior anti-PD-1 directed therapy (mAb or small molecule) are not eligible

Max Age: 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2024-12-29 (Actual); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Phase I: Recommended Phase II Dose (RP2D) | 60 days
  If one or fewer dose limiting toxicities (DLT's) occur in 6 participants the study will advance to the next dose level. If 2 or more DLT's occur at a dose level, the prior dose level will be identified as the RP2D.
Phase II: Rate of Continued Complete Remission (CR) | 1 year post surgery
  Continued complete remission by computed tomography (CT) scan 1 year after surgery.

SECONDARY OUTCOMES:
Percentage of Participants with Event Free Survival (EFS) | 1 year post surgery
  EFS: The time from diagnostic biopsy until the earliest of: death, local recurrence, new metastatic disease, progression of metastatic disease or secondary malignancy, or date of last contact.
Overall Survival (OS) Rate | 1 year post surgery
  The percentage of participants alive at 1 year post surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick A. Thompson, MD, Principal Investigator — University of North Carolina, Chapel Hill; Mihaela M Druta, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute, Coordinating Center
Locations (22):
- United States (22):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Los Angeles, USC Norris Comprehensive Cancer Center, Los Angeles, California
  - Children's Hospital of Colorado, Aurora, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I DuPont Hospital for Children, Wilmington, Delaware
  - Shand's Hospital for Children at the University of Florida, Gainesville, Florida
  - Nemours Children's Hospital, Jacksonville, Florida
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Nemours Children's Clinic, Orlando, Florida
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Coordinating Center, Tampa, Florida
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University, Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University of North Carolina at Chapel Hill, UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Carolina Medical Center, Levine Cancer Institute, Charlotte, North Carolina
  - Duke Health, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas